CLINICAL TRIAL: NCT04604522
Title: Evaluating Clonogenic Epithelial Cell Populations in Patients With Bronchiolitis Obliterans Syndrome
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2020-0325; NCI-2020-07790 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0325 (Other: M D Anderson Cancer Center); K23AI117024 (NIH)
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Bronchiolitis Obliterans
MeSH Terms: conditions — Bronchiolitis Obliterans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, airway brushings
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Ancillary-correlative (biospecimen collection, chart review): Patients undergo collection of blood samples and 6 brushings of the airway during SOC bronchoscopy. Patients' medical records are also reviewed for data collection.
  Interventions: Procedure: Biospecimen Collection; Other: Medical Chart Review

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood, airway brushings.
Other: Medical Chart Review — Patients' medical records are reviewed
  Other Names: Chart Review

SUMMARY:
This study investigates a type of cell, called abnormal clonogenic epithelial cells, in patients with bronchiolitis obliterans syndrome who have had an donor stem cell transplant or a lung transplant. Learning more about clonogenic cells in these patients may help doctors to detect signs of bronchiolitis obliterans syndrome earlier in future patients.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To characterize epithelial cell phenotypes in allogeneic hematopoietic cell transplant (allo-HCT) recipients at MD Anderson Cancer Center (MDACC) and in lung transplant recipients at Houston Methodist who have bronchiolitis obliterans syndrome (BOS).

OUTLINE:

Patients undergo collection of blood samples and 3 brushings of the airway during standard of care (SOC) bronchoscopy. After the bronchoscopy, patients undergo 2 nasal brushings (swabs). Patients' medical records are also reviewed for data collection.

After completion of study, patients are followed for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Allo-HCT recipients undergoing a bronchoscopy at MDACC who consent to undergoing study airway brushings in addition to clinically indicated bronchoscopic procedures (e.g. bronchoalveolar lavage)

  * 5 patients with advanced BOS - forced expiratory volume in one second (FEV1) =< 75% predicted and meeting other National Institutes of Health (NIH) criteria (FEV1/forced vital capacity [FVC] ratio 0.7, presence of air trapping or graft versus host disease [GVHD] of another organ)
  * 5 patient with early BOS - at least 10% decline in FEV1 from baseline values, with FEV1 >= 75% predicted, and 1 high-risk feature:

    * Active systemic chronic GVHD with new early airflow obstruction OR
    * Respiratory viral infection in last three months with resolution of viral symptoms but new airflow obstruction
  * 3 patients with no pulmonary impairment (FEV1 within 5% of baseline values)
* Lung allograft recipients undergoing a bronchoscopy at Houston Methodist who consent to undergoing study airway brushing sin addition to clinically indicated bronchoscopy procedures

  * 5 patients with BOS Stage 2 or higher (>= 35% decline in FEV1 from baseline values)
  * 5 patient with BOS Stage 0p or 1 (10-35% decline in FEV1 from baseline values)
  * 3 patients undergoing screening bronchoscopy without decline in FEV1
  * patients with undiagnosed lung cancer and chronic obstructive pulmonary disease diagnosed by pulmonary function testing (FEV1/FVC less than the lower limit of normal with >20 pack-year history of smoking)

Exclusion Criteria:

* Bronchoscopy performed on emergency basis for life-threatening issues as opposed to routine diagnostic testing
* Patient unwilling to give consent for study airway brushings

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with BOS who have undergone an allo-HCT or lung allograft.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2020-08-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of abnormal epithelial cells between patients with bronchiolitis obliterans syndrome and those without | Up to 1 year
  The relationship between the proportion of abnormal cells and degree of air trapping and lung abnormalities will be described through simple correlation. Exploration of non-linear relationships or rank-based summaries will be considered as appropriate.

SECONDARY OUTCOMES:
Comparison of epithelial cell populations in allogeneic hematopoietic cell transplant recipients and lung graft recipients | Up to 1 year
  The relationship between the proportion of abnormal cells and degree of air trapping and lung abnormalities will be described through simple correlation. Exploration of non-linear relationships or rank-based summaries will be considered as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Sheshadri, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org